CLINICAL TRIAL: NCT00105482
Title: Testing the Effectiveness of Low Dose Naltrexone for Smoking Cessation and Minimization of Post-cessation Weight Gain
Brief Title: Targeted Interventions for Weight-Concerned Smokers
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NIAAAOMA15632; P50AA015632 (NIH); 9P50AA015632 (NIH)
Record Dates: First submitted 2005-03-14; First posted 2005-03-15 (Estimated); Results first posted 2013-03-05 (Estimated); Last update posted 2013-03-05 (Estimated); Status verified 2013-01

CONDITIONS: Nicotine Dependence
Keywords: Tobacco; Smoking; Weight; Weight perception; Naltrexone
MeSH Terms: conditions — Tobacco Use Disorder; Smoking; Body Weight | interventions — Naltrexone; Behavior Therapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Naltrexone, Transdermal Nicotine (Experimental): Arm 1 (Experimental) = Transdermal nicotine replacement (21 mg for first 6 weeks post-quit then 14 mg for 2 weeks) once per day + Naltrexone 25 mg oral capsule once per day
  Interventions: Drug: Naltrexone; Drug: Transdermal nicotine replacement; Behavioral: Behavioral counseling
- Placebo Naltrexone, Transdermal Nicotine (Placebo Comparator): Arm 2 (Placebo Comparator) = Transdermal nicotine replacement (21 mg for first 6 weeks post-quit then 14 mg for 2 weeks) once per day + Placebo Naltrexone 25 mg oral capsule once per day
  Interventions: Drug: Transdermal nicotine replacement; Behavioral: Behavioral counseling

INTERVENTIONS:
Drug: Naltrexone — Drug: Naltrexone 12.5 mg oral capsule once per day for 1 day then 25 mg oral capsule once per day for 27 weeks
  Arms: Naltrexone, Transdermal Nicotine
Drug: Transdermal nicotine replacement — Transdermal nicotine replacement (21 mg for first 6 weeks post-quit then 14 mg for 2 weeks) once per day + naltrexone 25 mg oral capsule once per day
Behavioral: Behavioral counseling — Brief behavioral counseling and research assessments are provided for two sessions prior to the quit date and then weekly for two weeks, bi-weekly for a month and every four weeks thereafter.

SUMMARY:
Weight gain after quitting smoking is an important barrier to treatment for many smokers. This study will test a drug called naltrexone with weight-concerned smokers to investigate whether or not this drug both improves smoking cessation quit rates and minimizes post quit weight gain.

DETAILED DESCRIPTION:
This is a 6-month randomized, double-blind, placebo controlled trial of 25 mg naltrexone for smoking cessation in a sample of 270 male and female weight-concerned smokers. Participants also receive transdermal nicotine replacement therapy during the first 8 weeks of the study, which they begin on their quit date. Naltrexone study medication will be started a week before their quit date and continued through the six-month period. Brief behavioral counseling and research assessments are provided for two sessions prior to the quit date and then weekly for two weeks, bi-weekly for a month and every four weeks thereafter. A follow-up appointment is completed at 12 months after participants' quit date.

The primary outcomes are six-month point prevalence abstinence and post-cessation weight gain for those who are continuously abstinent (not even a puff).

Secondary outcomes include an examination of alcohol consumption, evaluation of urges, other measures of smoking cessation success, point prevalence abstinence at 12 months, and food preferences. A number of tertiary measures will be obtained for examining predictors of smoking cessation, weight gain, and naltrexone response.

ELIGIBILITY:
Inclusion Criteria:

* 1. Concern about gaining weight after quitting. This will be assessed using questionnaires that will provide a rating system to determine qualified participants.
* 2. Age 18 and older.
* 3. Willingness and ability to give written consent.
* 4. Smoking greater than 10 cigarettes per day for at least 1 year.
* 5. At least one prior attempt to stop smoking.
* 6. Baseline expired carbon-monoxide level of at least 10 ppm.
* 7. Weigh at least 100 lbs.
* 8. English speaking.
* 9. One person per household.

Exclusion Criteria:

* 1. Pregnant or nursing women or women attempting to conceive.
* 2. Unstable cardiac disease.
* 3. History of dermatoses.
* 4. Current alcohol or drug dependence other than nicotine dependence.
* 5. Serious current neurologic, psychiatric or medical illness, including those with a significant risk of committing suicide based on history or investigator's judgment.
* 6. Chronic pain conditions necessitating opioid treatment (naltrexone, an opioid antagonist, will make these medications ineffective).
* 7. History of cirrhosis or significant hepatocellular injury as evidenced by SGOT or SGPT >3 x normal or elevated bilirubin.
* 8. Current use of smokeless tobacco, pipes, cigars, nicotine gum, patch, nasal spray, inhaler, or lozenges.
* 9. Patients requiring concomitant therapy with any psychotropic drug or on any drug with a psychotropic component except those who are on a stable dose of an Selective Serotonin Reuptake Inhibitor for at least two months for the indications of Major Depressive Disorder, Premenstrual Syndrome (PMS) or Premenstrual Dysphoric Disorder (PMDD).
* 10. Subjects with a positive opiate urine drug screen will be excluded to avoid precipitating opiate withdrawal.
* 11. Current use of opiates.
* 12. Currently on a medically prescribed diet.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 172 (Actual)
Dates: Start 2005-01; Primary Completion 2009-04 (Actual); Study Completion 2009-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie O'Malley, PhD, Principal Investigator — Yale University
Locations (1):
- Yale University School of Medicine Substance Abuse Treatment Unit, New Haven, Connecticut, United States

REFERENCES:
- [Result] Toll BA, White M, Wu R, Meandzija B, Jatlow P, Makuch R, O'Malley SS. Low-dose naltrexone augmentation of nicotine replacement for smoking cessation with reduced weight gain: a randomized trial. Drug Alcohol Depend. 2010 Oct 1;111(3):200-6. doi: 10.1016/j.drugalcdep.2010.04.015. Epub 2010 Jun 12. PMID 20542391
- See also: This website describes the Transdisciplinary Tobacco Use Research Center at Yale University. Click here for more information about the study: Targeted Interventions for Weight-concerned Smokers. — http://www.quitwithyale.org

RESULTS

PARTICIPANT FLOW:
Groups:
- Naltrexone: Arm 1 (Experimental) = Transdermal nicotine replacement (21 mg for first 6 weeks post-quit then 14 mg for 2 weeks) once per day + Naltrexone 25 mg oral capsule once per day
  Transdermal nicotine replacement : Transdermal nicotine replacement (21 mg for first 6 weeks post-quit then 14 mg for 2 weeks) once per day + naltrexone 25 mg oral capsule once per day
  Naltrexone : Drug: Naltrexone 12.5 mg oral capsule once per day for 1 day then 25 mg oral capsule once per day for 27 weeks
  Behavioral counseling : Brief behavioral counseling and research assessments are provided for two sessions prior to the quit date and then weekly for two weeks, bi-weekly for a month and every four weeks thereafter.
- Placebo: Arm 2 (Placebo Comparator) = Transdermal nicotine replacement (21 mg for first 6 weeks post-quit then 14 mg for 2 weeks) once per day + Placebo Naltrexone 25 mg oral capsule once per day
  Behavioral counseling : Brief behavioral counseling and research assessments are provided for two sessions prior to the quit date and then weekly for two weeks, bi-weekly for a month and every four weeks thereafter.
Period: Overall Study
Arm/Group | Naltrexone | Placebo
Started | 87 | 85
Completed | 28 | 30
Not Completed | 59 | 55
Not completed — Adverse Event | 1 | 1
Not completed — Lost to Follow-up | 26 | 17
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Lost Interest | 29 | 32
Not completed — Scheduling Conflict | 2 | 3
Not completed — Withdrawn by PI | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Naltrexone | Placebo | Total
Number analyzed (Participants) | 87 | 85 | 172
Age Continuous [Mean (Standard Deviation); unit: years] | 43.2 (10.0) | 45.5 (11.3) | 44.4 (10.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 62 | 61 | 123
  Male | 25 | 24 | 49

OUTCOME MEASURES:

1. Primary Outcome: Weight Gain at 26 Weeks.
Description: Weight change from baseline measured at 26 weeks.
Time Frame: 26 weeks
Population: All patients who were randomized comprised the primary ITT population.
Measure: Mean (Standard Deviation); unit: pounds
Arm/Group | Naltrexone | Placebo
Number analyzed (Participants) | 87 | 85
pounds | 6.75 (8.94) | 9.71 (9.19)

2. Primary Outcome: Point Prevalence Smoking Abstinence at 26 Weeks.
Description: The number of people that were abstinent from cigarette smoking at 26 weeks.
Time Frame: 26 weeks
Population: All patients who were randomized comprised the primary ITT population.
Measure: Number; unit: participants
Arm/Group | Naltrexone | Placebo
Number analyzed (Participants) | 87 | 85
participants | 19 | 23

3. Secondary Outcome: Weight Gain at 6 Weeks.
Description: Weight change from baseline measured at 6 weeks.
Time Frame: 6 weeks
Population: All patients who were randomized comprised the primary ITT population.
Measure: Mean (Standard Deviation); unit: pounds
Arm/Group | Naltrexone | Placebo
Number analyzed (Participants) | 87 | 85
pounds | 2.53 (4.58) | 2.19 (4.20)

4. Secondary Outcome: Point Prevalence Smoking Abstinence at 6 Weeks
Description: The number of people that were abstinent from cigarette smoking at 6 weeks.
Time Frame: 6 weeks
Population: All patients who were randomized comprised the primary ITT population.
Measure: Number; unit: participants
Arm/Group | Naltrexone | Placebo
Number analyzed (Participants) | 87 | 85
participants | 33 | 43

5. Secondary Outcome: Cigarettes Smoked Per Day.
Description: Average number of cigarettes smoked per day at 26 weeks.
Time Frame: 26 weeks
Population: Patients were analyzed per protocol.
Measure: Mean (Standard Deviation); unit: number of cigarettes
Arm/Group | Naltrexone | Placebo
Number analyzed (Participants) | 67 | 67
number of cigarettes | 7.10 (8.43) | 7.85 (8.35)

ADVERSE EVENTS:
Time Frame: 26 months
Arm/Group | Naltrexone | Placebo
Serious Adverse Events (participants affected / at risk) | 2/87 | 2/85
Other Adverse Events (participants affected / at risk) | 51/87 | 51/85
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Naltrexone (N=87) | Placebo (N=85)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0) — Anxiety leading to hospitalization.
Abnormal EKG (Cardiac disorders) | 1 (1) | 0 (0) — Abnormal EKG leading to hospitalization.
Finger Laceration (General disorders) | 0 (0) | 1 (1) — Patient accidentally cut their finger with a saw, injury resulted in hospitalization.
Thyroid Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) — Patient was diagnosed with Thyroid Cancer.
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Naltrexone (N=87) | Placebo (N=85)
Abdominal Pain (General disorders) | 30 (30) | 24 (24)
Anxiety (Psychiatric disorders) | 39 (39) | 35 (35)
Blurred Vision (Eye disorders) | 10 (10) | 11 (11)
Constipation (Gastrointestinal disorders) | 29 (29) | 28 (28)
Decreased Appetite (Metabolism and nutrition disorders) | 43 (43) | 28 (28)
Depression (Psychiatric disorders) | 27 (27) | 31 (31)
Dizziness (Nervous system disorders) | 34 (34) | 25 (25)
Fatigue (General disorders) | 44 (44) | 37 (37)
Headache (Nervous system disorders) | 39 (39) | 36 (36)
Increased Appetite (Metabolism and nutrition disorders) | 43 (43) | 36 (36)
Increased Bowel Freq (Gastrointestinal disorders) | 11 (11) | 16 (16)
Insomnia (General disorders) | 40 (40) | 37 (37)
Itching (Skin and subcutaneous tissue disorders) | 31 (31) | 32 (32)
Change in Libido (General disorders) | 14 (14) | 13 (13)
Missed Period (Reproductive system and breast disorders) | 3 (3) | 2 (2)
Muscle Weakness (Musculoskeletal and connective tissue disorders) | 10 (10) | 13 (13)
Nausea (Gastrointestinal disorders) | 48 (48) | 25 (25)
Rapid Heartbeat (Cardiac disorders) | 18 (18) | 19 (19)
Rash (Skin and subcutaneous tissue disorders) | 24 (24) | 26 (26)
Sleepiness (General disorders) | 33 (33) | 23 (23)
Sweating (Endocrine disorders) | 40 (40) | 21 (21)
Vivid Dreams (Psychiatric disorders) | 51 (51) | 51 (51)
Vomiting (Gastrointestinal disorders) | 19 (19) | 4 (4)
Other (General disorders) | 31 (31) | 28 (28)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes